CLINICAL TRIAL: NCT00325416
Title: A Study of Intensive-Dose Melphalan and Topotecan (MT) Followed by Autologous Stem Cell Rescue in Patients With Multiple Myeloma.
Brief Title: Study of Melphalan and Topotecan (MT) Followed by Autologous Stem Cell Rescue in Patients With Multiple Myeloma.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: GlaxoSmithKline (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12733
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Multiple Myeloma
Keywords: melphalan; topotecan; topoisomerase; bone marrow transplant; drug sequence
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Topotecan; Bone Marrow Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Age Group A - Melphalan and Topotecan plus Stem Cell Rescue (Experimental): Participants 18 - 60 years of age. Intensive-Dose Melphalan and Topotecan (MT) followed by Stem Cell transplant.
  Interventions: Drug: melphalan; Drug: topotecan (TPT); Procedure: Autologous Stem Cell Rescue
- Age Group B - Melphalan and Topotecan plus Stem Cell Rescue (Active Comparator): Participants 61 years of age or older. Intensive-Dose Melphalan and Topotecan (MT) followed by Stem Cell transplant.
  Interventions: Drug: melphalan; Drug: topotecan (TPT); Procedure: Autologous Stem Cell Rescue

INTERVENTIONS:
Drug: melphalan — (Days -4,-3,-2) 50 mg/m^2/day IV over 30 minutes (total dose 150 mg/m^2)
  Other Names: Alkeran®
Drug: topotecan (TPT) — Phase I Dose Escalation: Level 1 - 20 mg/m^2; Level 2 - 30 mg/m^2; Level 4 - 54 mg/m^2; Level 5 - 72 mg/m^2; Level 6 - 96 mg/m^2; Level 7 - 127.8 mg/m^2; Level 8 - 170.1 mg/m^2
  Phase II: Treatment at maximum tolerated dose (MTD)
  Other Names: Hycamtin®
Procedure: Autologous Stem Cell Rescue — Day 0
  Other Names: Bone Marrow Transplant; Stem Cell Transplant

SUMMARY:
The purpose of this research study is to determine the safest dose of topotecan when given in a high dose before a stem cell transplant; topotecan will be given with melphalan.

DETAILED DESCRIPTION:
The stem cells being transplanted are cells found in the bone marrow and blood that are responsible for making red blood cells, white blood cells, and platelets. The stem cells are collected by a process called leukapheresis and will be frozen for later use. After receiving the chemotherapy drugs, the stem cells will be thawed and given like a blood transfusion. This is called autologous stem cell transplant or rescue. The study doctors will be measuring how well the disease responds to the drugs as well as any side effects to the drugs. During the course of this study, blood and bone marrow samples will be obtained to measure levels of the chemotherapy drugs as well as levels of certain enzymes (proteins).

The staff of the Blood and Marrow Transplant program will continue to collect information about the participant's disease and its treatment for the rest of their life.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma Criteria = Newly diagnosed with drug sensitive disease (>50% tumor response to standard chemotherapy) and poor prognostic indicators, such as Salmon-Durie stage III, serum b-2-microglobulin >3.0 mg/L, high proliferative fraction or hypodiploidy. Relapsed patients after a response to standard chemotherapy. Patients with primary refractory disease. Patients with non-secretory multiple myeloma are eligible for enrollment on this study. They will be followed for toxicity, survival and molecular endpoint analyses, but will not be followed for response. Patients with plasma cell leukemia, either occurring de novo or arising from existing multiple myeloma, are ineligible for this study.
* Patients greater than or equal to 18 years of age are eligible.
* Patients must have histologically confirmed diagnosis by a pathologic review at the H. Lee Moffitt Cancer Center and Research Institute.
* Patients must have undergone a complete psychosocial evaluation and been considered capable of compliance.
* Patients willing and able to receive palifermin (young cohort only)

Exclusion Criteria:

* Patients with a diffusing lung capacity oxygenation (DLCO) less than 50% (adjusted) of normal or with symptomatic obstructive or restrictive disease are ineligible.
* Patients with a serum creatinine of greater than 2.0 mg/dL OR a creatinine clearance of less than 40 ml/minute. Creatinine clearance can be measured or calculated. Patients with renal dysfunction secondary to multiple myeloma may be enrolled at the discretion of the principal investigator. However, patients on hemodialysis or peritoneal dialysis are ineligible.
* Patients with a total bilirubin greater than 2.0 mg/dL and serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) greater than two and a half times normal (unless due to primary malignancy), or a history of severe hepatic dysfunction are ineligible.
* Patients who have evidence of severe cardiac dysfunction are ineligible. A gated blood pool (MUGA) scan must show an ejection fraction of at least 50%. Patients must be free of major heart disease. Patients are ineligible if they have received a total dose of doxorubicin of greater than 450 mg/m2 (or daunorubicin equivalent) unless the left ventricular ejection fraction by MUGA scan is at least 50%. Patients must not be taking nitroglycerin preparations for angina pectoris or antiarrhythmic drugs for major ventricular dysrhythmias. Patients with essential hypertension controlled with medications are eligible for study. Any patient with congenital or acquired heart disease or cardiac arrhythmias will have a cardiology consult and evaluation.
* Patients with active infections are ineligible.
* Patients who are HIV antibody positive are ineligible.
* Patients with active leptomeningeal involvement are ineligible. Patients with a history of previous cerebrospinal fluid (CSF) tumor involvement without symptoms or signs are eligible provided the CSF is now free of disease on lumbar puncture and MRI of the brain shows no tumor involvement. Patients with severe symptomatic central nervous system (CNS) disease of any etiology are ineligible.
* Patients with uncontrolled insulin-dependent diabetes mellitus or uncompensated major thyroid or adrenal dysfunction are ineligible.
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of > or = 2 are ineligible. Patients with ECOG performance status 2 to 3 secondary to bone pain may be enrolled at the discretion of the institutional investigator. Patients with ECOG performance status 2 to 3 secondary to a potentially reversible disease-related problem may be enrolled at the discretion of the institutional investigator.
* Patients who are pregnant or lactating are ineligible.
* Patients with any previous malignancy other than non-melanoma skin cancer are ineligible, unless the patient is without evidence of disease > or = 5 years after the treatment for the cancer was completed.
* Patients previously treated with topotecan or any other topoisomerase I inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2001-11-19 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Sullivan, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: H. Lee Moffitt Cancer Center & Research Institute — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I: 129 (70 Group A and 60 Group B) participants were enrolled during the Phase I portion.
  Phase II: 48 (40 Group A and 8 Group B) participants were enrolled during the Phase II portion.
  Both Phases: 72 Phase I participants were still on study when Phase II began.
Groups:
- Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue: Participants 18 - 60 years of age. Intensive-Dose Melphalan and Topotecan (MT) followed by Stem Cell transplant.
  melphalan: (Days -4,-3,-2) 50 mg/m^2/day IV over 30 minutes (total dose 150 mg/m^2)
  topotecan (TPT): Phase I Dose Escalation: Level 1 - 20 mg/m^2; Level 2 - 30 mg/m^2; Level 4 - 54 mg/m^2; Level 5 - 72 mg/m^2; Level 6 - 96 mg/m^2; Level 7 - 127.8 mg/m^2; Level 8 - 170.1 mg/m^2
  Phase II: Treatment at maximum tolerated dose (MTD)
  Autologous Stem Cell Rescue: Day 0
- Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue: Participants 61 years of age or older. Intensive-Dose Melphalan and Topotecan (MT) followed by Stem Cell transplant.
  melphalan: (Days -4,-3,-2) 50 mg/m^2/day IV over 30 minutes (total dose 150 mg/m^2)
  topotecan (TPT): Phase I Dose Escalation: Level 1 - 20 mg/m^2; Level 2 - 30 mg/m^2; Level 4 - 54 mg/m^2; Level 5 - 72 mg/m^2; Level 6 - 96 mg/m^2; Level 7 - 127.8 mg/m^2; Level 8 - 170.1 mg/m^2
  Phase II: Treatment at maximum tolerated dose (MTD)
  Autologous Stem Cell Rescue: Day 0
Period: Phase I: Dose Escalation
Arm/Group | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue
Started | 70 | 60
Completed | 48 | 44
Not Completed | 22 | 16
Not completed — Pre-transplant screen failure | 8 | 9
Not completed — Denial of insurance coverage | 7 | 4
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Inability to collect adequate stem cells | 0 | 1
Period: Phase II: Treatment at MTD
Arm/Group | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue
Started | 78 | 42
Proceeded From Phase I to Phase II | 38 | 34
Enrolled During Phase II | 40 | 8
Completed | 78 | 40
Not Completed | 0 | 2
Not completed — denial of insurance coverage | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants: 177 included in Baseline; 129 included in Phase I Maximum Tolerated Dose Outcome; 51 Phase II participants with responsive disease prior to transplant were re-evaluated for the Overall Response Rate; 79 treated in Phase II and evaluable at time of analysis are included in the Event Free Survival and Overall Survival Outcome Measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue | Total
Number analyzed (Participants) | 109 | 68 | 177
Age, Continuous [Median (Full Range); unit: years] | 46 [32 to 60] | 68.5 [61 to 76] | 54 [32 to 76]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 10 | 119
  >=65 years | 0 | 58 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 29 | 68
  Male | 70 | 39 | 109
Region of Enrollment [Number; unit: participants]
  United States | 109 | 68 | 177

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Maximum Tolerated Dose (MTD) Level
Description: MTD of topotecan in multiple myeloma patients receiving autologous transplant when give with melphalan 150 mg/m^2 for three days. Two parallel dose escalations were used, one each for young (18-60 years of age) and elderly patients (> 61 years of age). Elderly patients began a dose level once it had been found to be safe for the young cohort. The purpose of this approach was to expand the access of this trial to elderly patients while ensuring safety.
  Phase I Dose Escalation: Level 1 - 20 mg/m^2; Level 2 - 30 mg/m^2; Level 4 - 54 mg/m^2; Level 5 - 72 mg/m^2; Level 6 - 96 mg/m^2; Level 7 - 127.8 mg/m^2; Level 8 - 170.1 mg/m^2
Time Frame: Phase I - 5 years, 2 months
Population: Phase I Dose Escalation participants.
Measure: Number; unit: mg/m^2
Arm/Group | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue
Number analyzed (Participants) | 69 | 60
mg/m^2 | 127.8 | 30

2. Primary Outcome: Phase II Participants - Overall Response Rate
Description: Re-evaluation of participants who had responsive disease prior to transplant. All changes in monoclonal protein and immunoglobulins will be referenced to those levels obtained immediately prior to cyclophosphamide priming chemotherapy. Complete Response (CR): A CR will be defined as the disappearance of the monoclonal protein by immunofixation studies of serum and urine (100x concentrate) and less than or equal to 5% plasma cells in a bone marrow aspirate. Partial Response (PR): 50% - 74% decrease in the measurable monoclonal protein (M-component from an SPEP and/or UPEP with immunofixation).
Time Frame: Phase II - Phase start at 62 months up to 120 months
Population: Phase II (treatment at MTD) participants with responsive disease prior to transplant.
Measure: Number; unit: percentage of participants
Arm/Group | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue
Number analyzed (Participants) | 23 | 28
percentage of participants
  Overall Response Rate | 65 | 57
  Complete Response Rate | 26 | 18
  Partial Response Rate | 39 | 39

3. Secondary Outcome: Phase II Event Free Survival (EFS)
Description: Time to treatment failure, which is defined as the time from day 0 to the time of progressive disease. Progressive disease is defined by unequivocal objective evidence and constitutes any of the following: 1). an increase in the total amount of monoclonal protein (M-component from Serum Protein Electrophoresis (SPEP) and/or Urine Protein Electrophoresis (UPEP) with immunofixation) by more than 100% from the lowest level of serum myeloma protein seen after high-dose chemotherapy by serum protein electrophoresis; 2). an increase in the total amount of monoclonal protein above the remission level of the myeloma peak (i.e., an increase of >25% above the lowest level in a 24 hour urine or serum protein; 3). the reappearance of the M-protein if the patient had entered a CR: 4). definite increase in the size (> 1 cm) or number of lytic bone lesions. Compression fractures do not constitute a relapse.
Time Frame: Phase II - Phase start at 62 months up to 120 months
Population: Phase II (treatment at MTD) evaluable participants at time of analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue
Number analyzed (Participants) | 39 | 40
months | 13.3 [11.6 to 21.5] | 21.3 [14.9 to 27.2]

4. Secondary Outcome: Phase II Overall Survival (OS)
Description: Time from start of treatment until death from any cause.
Time Frame: Phase II - Phase start at 62 months up to 120 months
Population: Phase II (treatment at MTD) evaluable participants at time of analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue
Number analyzed (Participants) | 39 | 40
months | 63 [35 to NA] — not yet reached | 62 [45 to NA] — not yet reached

5. Other Pre Specified Outcome: Pharmacokinetic Profiles of High Dose Topotecan and Melphalan
Description: Evaluate the pharmacokinetic profiles of high dose topotecan and melphalan and to investigate the pharmacodynamic relationships with respect to the efficacy and toxicity of this regimen in each age group. Pharmacokinetics of Topotecan: For all dose levels, topotecan levels on Day -4 will be obtained at -15 min, 20 min into 30 min infusion, and 5 min, 15 min, 30 min, 1 h, 2 h, 4 h, 8 h, and 23 h after the 30 min infusion. Pharmacokinetics of Melphalan: For all dose levels, melphalan levels during the first day of cytoxan priming chemotherapy and on Day -4 will be obtained before, at the end of the infusion, and 5 minutes (min), 15 min, 30 min, 45 min, 60 min, 90 min, 120 min and 180 min after the infusion. The infusion time for the test dose of melphalan is over 5 min and for the high-dose is over 30 min.
Time Frame: Predetermined time points in protocol
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Amount, Activity and Subcellular Distribution of Topoisomerase I With Clinical Response and Toxicity
Description: Laboratory Correlates will be summarized using descriptive statistics.
Time Frame: Laboratory study (no specific time points)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: DNA Topoisomerase I Amount, Activity, or Subcellular Distribution
Description: Laboratory Correlates will be summarized using descriptive statistics.
Time Frame: Laboratory study (N/A)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Genomic DNA Sequence Variations and Correlate With Toxicity to Melphalan and Topotecan
Description: Laboratory Correlates will be summarized using descriptive statistics.
Time Frame: Laboratory study (N/A)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Breast Cancer Resistance Protein (BCRP) Expression
Description: BCRP function will be assayed in multiple myeloma patient bone marrow aspirates obtained before and during high dose chemotherapy. BCRP function is expressed as the change in relative fluorescence in topotecan versus control cells. The distribution of paired differences in BCRP, a continuous variable, will be summarized using descriptive statistics and will be correlated with response and toxicity.
Time Frame: Laboratory study (N/A)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 years
Arm/Group | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue
Serious Adverse Events (participants affected / at risk) | 27/109 | 23/68
Other Adverse Events (participants affected / at risk) | 0/109 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age Group A - Melphalan and Topotecan Plus Stem Cell Rescue (N=109) | Age Group B - Melphalan and Topotecan Plus Stem Cell Rescue (N=68)
Neutrophils/granulocytes - low (Blood and lymphatic system disorders) | 1 | 1
Platelets - low (Blood and lymphatic system disorders) | 1 | 1
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 2 | 0
Fever (in the absence of neutropenia) (General disorders) | 11 | 7
Diarrhea (Gastrointestinal disorders) | 4 | 1
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Infection - Other - cellulitis (Infections and infestations) | 1 | 0
ALT, SGPT 9serum glutamic pyruvic transaminase) - increased (Metabolism and nutrition disorders) | 1 | 0
AST, SGOT (serum glutamic oxaloacetic transaminase) - increased (Metabolism and nutrition disorders) | 1 | 0
Alkaline phosphatase - increased (Metabolism and nutrition disorders) | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal/Soft Tissue - Other - Knee (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal/Soft Tissue - Other - Rotator cuff (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathy: motor (Nervous system disorders) | 1 | 0
Neuropathy: sensory (Nervous system disorders) | 2 | 0
Pain - Back (General disorders) | 2 | 1
Pain - Bone (General disorders) | 2 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0
Hypertension (Cardiac disorders) | 1 | 2
Blurred vision (Ear and labyrinth disorders) | 0 | 1
Eye - NOS (visual changes) (Eye disorders) | 1 | 0
Fatigue (General disorders) | 3 | 0
Febrile neutropenia (Infections and infestations) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Symptomatic pericarditis (Cardiac disorders) | 1 | 0
Edema: limb (Blood and lymphatic system disorders) | 1 | 0
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Infection: Catheter related (Infections and infestations) | 2 | 2
Hypotension (Cardiac disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1
Pain - Chest wall (General disorders) | 5 | 1
Infection - Other - Sepsis syndrome (Infections and infestations) | 1 | 0
Rigors/chills (General disorders) | 3 | 2
Hallucinations (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hemoglobin - low (Blood and lymphatic system disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 2 | 2
Infection - Lung (pneumonia) (Infections and infestations) | 4 | 0
Pain - Head/headache (General disorders) | 4 | 0
Infections and infestations - Other - Herpes Zoster (Infections and infestations) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dehydration (Gastrointestinal disorders) | 0 | 2
Infection- Other - CMV Viremia (Infections and infestations) | 0 | 1
Infection - Other - Residual enteritis (Infections and infestations) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0
Pain - Extremity - limb (General disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Pain - Chest/thorax NOS (General disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 1
Flushing (Vascular disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Renal and urinary disorders - Other - decreased urine output (Renal and urinary disorders) | 0 | 2
Infection - Rectum (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Psychiatric disorders - Other - mental status change (Psychiatric disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Creatinine - high (Renal and urinary disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Infection - Sinus (Infections and infestations) | 0 | 1
Wound (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 0
Death, NOS (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Data on presence of chromosomal abnormalities at time of diagnosis were not available for majority of patients. The cancer center will continue to collect information about the participant's disease and its treatment for the rest of their life.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes